CLINICAL TRIAL: NCT02855450
Title: An 8 Week Phase Ib, Monocentric, Randomized, Double-masked, Parallel Groups, Study With a 24 Week Follow-up to Evaluate Safety and Potential Efficacy of a 180 μg/ml rhNGF Eye Drops Solution Vs Vehicle in Patients With Glaucoma
Brief Title: Study to Evaluate Safety and Efficacy of rhNGF Eye Drops Solution Versus Vehicle in Patients With Glaucoma
Acronym: NGF-Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NGF0314
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — cenegermin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rhNGF (Experimental): rhNGF (Recombinant Human Nerve Growth Factor) 180 μg/ml eye drops solution
  Interventions: Drug: rhNGF
- Vehicle (Placebo Comparator): Ophthalmic Placebo solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: rhNGF — Recombinant Human Nerve Growth Factor 180μg/ml (one 35 μl drop equals to 6.30 μg of rhNGF) reconstituted solution three times a day (TID) for 8 weeks of treatment.
  Other Names: cenegermin
  Arms: rhNGF
Drug: Vehicle — Ophthalmic Placebo solution of the same composition as the test product with the exception of rhNGF reconstituted solution times a day (TID) for 8 weeks of treatment.
  Other Names: placebo
  Arms: Vehicle

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of a 180μg/ml TID dose regimen of recombinant human nerve growth factor (rhNGF) eye drop solution administered over 8 weeks versus a vehicle control in patients with progressive primary open-angle glaucoma despite IOP control.

The secondary objectives are to measure the changes in BCDVA, visual field, ERG and structural changes in ganglion cell layer and nerve fiber layer thickness measured by optical coherence tomography. The secondary outcomes will be examined at 1, 4 and 8 weeks of therapy, and at 4 and 24 weeks after cessation of therapy (Week 12 visit and Week 32 visit), and will include functional assessments to investigate evidence of a persistent biological effect after discontinuation of the study treatment.

DETAILED DESCRIPTION:
This is an 8 Week phase Ib, monocentric, randomized, double-masked, vehicle controlled, parallel groups, study with a 24 Week follow-up period to evaluate the safety and potential efficacy of a 180 μg/ml recombinant human nerve growth factor (rhNGF) eye drops solution versus vehicle in 60 study participants with chronic primary open angle glaucoma.

Participants may qualify with either progressive optic neuropathy despite maximal current therapy (i.e. IOP reduction), or with stabilized IOP but diminished vision (central or peripheral).

Participants with a qualifying eye will be randomized 2:1 to topical recombinant human nerve growth factor (rhNGF) therapy or vehicle placebo control. Examinations for safety and efficacy will occur one week following initiation of therapy, and at 4, 8, 12 and 32 weeks.

All participants in either arm will be followed clinically at 4 weeks after cessation of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older. Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.
2. Participant's clinical diagnosis must be consistent with glaucoma characterized by the following features: a) clinical evidence of progressive RGC dysfunction and degeneration using visual field and/or a structural modality. There must be at least 3 reliable visual fields within 14 months prior to entering into the study; b) residual visual field preservation in at least 1 quadrant.
3. Participant must be medically able to undergo the testing required in the flowsheet of exam procedures.
4. Females of childbearing potential must agree to use an effective form of birth control.

Exclusion Criteria:

1. Participant has another optic nerve or retinal degenerative disease or co-morbidity causing significant vision loss, irrespective of whether it is currently treated or untreated, that could limit the possibility of visual recovery.
2. Participant is blind in one eye.
3. Participant has a requirement of acyclovir and/or related products during study duration. 4- Participant has evidence of corneal opacification or lack of optical clarity.
4. Participant has evidence of corneal opacification or lack of optical clarity.
5. Participant has undergone lens removal in the last 3 months, with or without intra-ocular lens implantation, or has undergone intra-ocular lens replacement within 3 months, or has undergone any other ocular surgery within 9 months prior to initiation of study drug.
6. Participant is receiving systemic steroids or other immunosuppressive medications.
7. Participant is currently participating in or has within the last 3 months participated in any other clinical trial of a non-clinically approved drug by ocular or systemic administration.
8. Participant has uveitis or other ocular inflammatory disease.
9. Participant has diabetic macular edema.
10. Participant has a history of ocular herpes zoster.
11. Participant is on chemotherapy.
12. Participant has a history of malignancy, not counting basal cell carcinomas, UNLESS it was treated successfully 2 years prior to inclusion in the trial.
13. Known hypersensitivity to one of the components of the study or procedural medications.
14. History of drug, medication or alcohol abuse or addiction.
15. Females of childbearing potential (those who are not surgically sterilized or post- menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

    1. are currently pregnant or,
    2. have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
    3. intend to become pregnant during the study treatment period or,
    4. are breast-feeding or,
    5. not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or IUD during the entire course of and 30 days after the study treatment periods.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD, PhD, Principal Investigator — , MD, PhD
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beykin G, Stell L, Halim MS, Nunez M, Popova L, Nguyen BT, Groth SL, Dennis A, Li Z, Atkins M, Khavari T, Wang SY, Chang R, Fisher AC, Sepah YJ, Goldberg JL. Phase 1b Randomized Controlled Study of Short Course Topical Recombinant Human Nerve Growth Factor (rhNGF) for Neuroenhancement in Glaucoma: Safety, Tolerability, and Efficacy Measure Outcomes. Am J Ophthalmol. 2022 Feb;234:223-234. doi: 10.1016/j.ajo.2021.11.002. Epub 2021 Nov 13. PMID 34780798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rhNGF | Vehicle
Started | 40 | 20
Completed | 35 | 20
Not Completed | 5 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set (SAF) The SAF includes all randomized subjects who received at least one dose of study medication. This safety population is used in the analysis of all safety endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF | Vehicle | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 25 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (13.98) | 62.2 (13.28) | 66.1 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 26 | 11 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 38 | 19 | 57
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Events as of Primary Safety Outcomes
Description: Unexpected Severe Progression Of Optic Neuropathy (USPON) is a composed parameter which required at least 28 single evaluations; it occurred if the subject answered Yes to any of the following 4 questions on unexpected severe progression:
  * Best Corrected Distance Visual Acuity (BCDVA): 'Yes' for at least one treated eye at any Follow-Up Visit after first study drug dose
  * Humphrey Visual Field (HVF): 'Yes' for at least one treated eye in at least one assessment during treatment or follow-up period
  * Electroretinography (ERG): 'Yes' for at least one treated eye at any Follow-Up Visit after first study drug dose
  * Optical Coherence tomography (OCT): 'Yes' for at least one treated eye at any Follow-Up Visit after first study drug dose
  Intolerance and allergy to the drug was identified based on preferred term of treatment-emergent adverse events.
  URAEs are unexpected related AE affecting ocular function. Local/systemic toxicities were identified via the AE form
Time Frame: At day 56/end of treatment
Population: Safety Set (SAF). The Safety Set includes all randomized subjects who received at least one dose of study medication. This safety population is used in the analysis of all safety endpoints. All analyses based on the SAF are summarized by the treatment received
Measure: Number; unit: Number of events
Arm/Group | rhNGF | Vehicle
Number analyzed (Participants) | 40 | 20
Number of events
  USPON | 0 | 2
  USPON during treatment period | 0 | 0
  Intolerance to the drug | 6 | 0
  Ocular URAEs | 1 | 1
  Local/systemic toxicities | 0 | 0

2. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Ocular Tolerability Score
Description: A ocular tolerability score was determined using a 100 mm VAS on which 0 meant No symptoms and 100 meant the Worst possible discomfort. The patients subjectively evaluated their ocular symptoms (foreign body sensation, burning or stinging, itching, pain, sticky feeling, blurred vision and photophobia) using the VAS giving the value they were feeling from none to an extreme value.
  The ocular symptoms were evaluated by the patients through the scale. Only "overall" values for primary eye and secondary eye are reported here under.
  An eye was considered as Primary eye, if
  * the eye was treated and
  * the investigator considered this eye as qualifying eye.
  * If both eyes were considered as qualifying eye, the right eye was chosen.
  The other eye was then considered as Secondary eye, if the eye was treated.
Time Frame: Change from baseline to days 7, 28 and 56 (Treatment period), and Day 84 (Follow up)
Population: The Safety Set includes all randomized subjects who received at least one dose of study medication. This safety population is used in the analysis of all safety endpoints. All analyses based on the SAF are summarized by the treatment received.
  Please note that there were major protocol deviations, so that no complete VAS data was reported during treatment period; for this reason the numbers of participants analyzed per row may differ from the Overall Numbers of Participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF | Vehicle
Number analyzed (Participants) | 40 | 20
score on a scale
  Day 7 - primary eye: number analyzed (Participants) | 34 | 18
  Day 7 - primary eye | 2.8 (9.09) | -2.1 (5.95)
  Day 28 - primary eye: number analyzed (Participants) | 36 | 16
  Day 28 - primary eye | 4.0 (11.22) | 1.0 (11.85)
  Day 56 - primary eye: number analyzed (Participants) | 32 | 16
  Day 56 - primary eye | 3.6 (16.08) | -0.9 (6.51)
  Day 84 - primary eye: number analyzed (Participants) | 32 | 17
  Day 84 - primary eye | -0.3 (11.81) | 0.3 (6.78)
  Day 7 - secondary eye: number analyzed (Participants) | 34 | 17
  Day 7 - secondary eye | 2.1 (9.44) | -1.4 (6.45)
  Day 28 - secondary eye: number analyzed (Participants) | 35 | 15
  Day 28 - secondary eye | 4.6 (13.25) | 1.2 (12.16)
  Day 56 - secondary eye: number analyzed (Participants) | 32 | 15
  Day 56 - secondary eye | 4.5 (16.64) | 0.6 (10.60)
  Day 84 - secondary eye: number analyzed (Participants) | 31 | 16
  Day 84 - secondary eye | -0.7 (12.95) | 1.5 (10.71)
Statistical Analysis 1: Comparison: rhNGF vs Vehicle; These statistics refer to Day 7 and primary eye; Test type: Superiority; p = 0.040, ANCOVA; Analysis results are obtained from an ANCOVA with treatment as factor and baseline value as covariate; Least square means difference = 4.7, 95% CI 2-sided [0.2 to 9.2]
Statistical Analysis 2: Comparison: rhNGF vs Vehicle; These statistics refer to Day 28 and primary eye; Test type: Superiority; p = 0.457, ANCOVA — Analysis results are obtained from an ANCOVA with treatment as factor and baseline value as covariate; least square mean difference = 2.4, 95% CI 2-sided [-4.1 to 9.0]
Statistical Analysis 3: Comparison: rhNGF vs Vehicle; These statistics refer to Day 56 and primary eye; Test type: Superiority; p = 0.283, ANCOVA — Analysis results are obtained from an ANCOVA with treatment as factor and baseline value as covariate; least square mean difference = 4.0, 95% CI 2-sided [-3.5 to 11.5]
Statistical Analysis 4: Comparison: rhNGF vs Vehicle; These statistics refer to Day 7 and secondary eye; Test type: Superiority — Analysis results are obtained from an ANCOVA with treatment as factor and baseline value as covariate; p = 0.147, ANCOVA; Least square means difference = 3.5, 95% CI 2-sided [-1.3 to 8.3]
Statistical Analysis 5: Comparison: rhNGF vs Vehicle; These statistics refer to Day 28 and secondary eye; Test type: Superiority — Analysis results are obtained from an ANCOVA with treatment as factor and baseline value as covariate; p = 0.421, ANCOVA; least square mean difference = 3.0, 95% CI 2-sided [-4.4 to 10.4]
Statistical Analysis 6: Comparison: rhNGF vs Vehicle; These statistics refer to Day 56 and secondary eye; Test type: Superiority — Analysis results are obtained from an ANCOVA with treatment as factor and baseline value as covariate; p = 0.327, ANCOVA; least square mean difference = 4.3, 95% CI 2-sided [-4.4 to 13.0]

ADVERSE EVENTS:
Time Frame: Treatment period: Day 0 (Therapy initiation), Day 7, Day 28, Day 56; Follow-up: Day 84, Day 224
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that started on or after the date of the First Study Treatment Administration. An AE was considered as TEAE if the Electronic Case Report Form question 'Did the event occurred:' was answered either with 'During Treatment Period' or 'During Follow-Up Period'.
Arm/Group | rhNGF | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/40 | 2/20
Other Adverse Events (participants affected / at risk) | 31/40 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF (N=40) | Vehicle (N=20)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF (N=40) | Vehicle (N=20)
Eye pain (Eye disorders) | 21 (26) | 2 (2)
Eye irritation (Eye disorders) | 6 (7) | 3 (3)
Photophobia (Eye disorders) | 8 (8) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 3 (4) | 1 (1)
Blepharitis (Eye disorders) | 3 (3) | 1 (1)
Vision blurred (Eye disorders) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 1 (1)
Lacrimation increased (Eye disorders) | 2 (2) | 1 (1)
Uveitis (Eye disorders) | 2 (2) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1)
Blepharochalasis (Eye disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival oedema (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Eyelid pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Meibonian gland dysfunction (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Haedache (Nervous system disorders) | 4 (4) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (3) | 1 (1)
Intraocular pressure test abnormal (Investigations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Loer respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 1 (2)
Photocoagulation (Surgical and medical procedures) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT02855450/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT02855450/SAP_001.pdf